CLINICAL TRIAL: NCT06907134
Title: A Controlled Trial of Smartphone-delivered Cognitive Behavioral Therapy for Adults Treated With Medication for Depressive Symptoms
Brief Title: The Purpose of the Study is to Investigate if a Smartphone App Combined With Internet Based Cognitive Behavioural Therapy (ICBT) Leads to Improved Symtoms in Depressive Adults on Antidepressive Medicine, Compared to a Wait-list Control Condition
Acronym: FIG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, PhD, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIG
Record Dates: First submitted 2024-12-20; First posted 2025-04-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Depressive Symptoms
Keywords: depressive symtoms; smartphone app; mobile game; internet-based cognitive behavioural therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: After the recruitment is finished, participants will be randomized to either ICBT treatment combined with a smartphone app or wait-list control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone delivered Internet-based Cognitive Behavioural Therapy (Experimental): The treatment consist of a 9 week long ICBT intervention based on an smartphone app with therapist support on demand.
  Interventions: Behavioral: Smartphone delivered internet-based Cognitive Behavioural Therapy
- No Intervention: Wait-list control condition (No Intervention): Wait-list control condition, participants have the option to contact the treatment team in case of worsened symptoms.

INTERVENTIONS:
Behavioral: Smartphone delivered internet-based Cognitive Behavioural Therapy — The intervention is 9 week long were partipants use an smartphone app based on CBT-principles with while having access to an internet platform where extra working material and therapist support is available on demand.
  Arms: Smartphone delivered Internet-based Cognitive Behavioural Therapy

SUMMARY:
The purpose of the study is to investigate if a smartphone app combined with internet delivered cognitive behavioural therapy (ICBT) leads to improved symptoms in depressive adults on antidepressive mediation. The participants in the treatment group will get access to a smartphone app based on CBT-principles for 9 weeks. They will also get access to an internet platform with extra treatment material based on CBT and receive therapist support on demand. Participants will be recruited in Sweden with nationwide recruitment.

DETAILED DESCRIPTION:
This study is a randomized controlled trial with the aim to investigate if an smartphone app in combination with ICBT can help adults (+18) on antidepressant medication who still suffers from depressive symptoms. Participants will either be randomized to a treatment phase for 9 weeks or to a wait-list control. The treatment primarily contains the installation and usage of a smartphone app where the participants can engage in a serious mobile game based on CBT-principles. They will receive access to a secure internet platform where they can find general guidelines about the app, and extra treatment modules (to use if needed). They will receive support on demand from a therapist during the whole treatment period.

Primary outcome measure is depressive symptoms (measured on the MADRAS scale). Secondary outcome measures will include measures of anxiety and quality of life. Pre-treatment measurement, post-treatment measurement, weekly measure, and 24 & 36 months follow up is planned to be collected through an online survey.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing drug treatment with an antidepressant mediated by an established care contact in (primary) care.
* 18 years or older.
* Be able to speak, read and write Swedish.
* Have access to a computer, tablet or other device with internet connection and smartphone to download the app.

Exclusion Criteria:

* Severe psychiatric or somatic problems that make participation difficult or impossible
* Ongoing abuse (via Audit and during interview)
* Acute suicidality
* Other ongoing psychological treatment or planned investigation.
* Planned dose change of medicine or change of medicine during pre-measurement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-02 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Ranging Scale (MADRS) | From enrollment to end of treament at 9 weeks. Follow-ups at 24 and 36 months after end of treatment.
  MADRS-S is a questionnaire including nine questions about depressive mental states. The questions aslo address experienced worry, ability to concentrate and initiative. Each question gives between 0 and 6 points. Maximum score is 54 points. Higher scores indicate higher levels of depression.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 | From enrollment to end of treament at 9 weeks. Follow-ups at 24 and 36 months after end of treatment.
  Measures symptoms of anxiety. 7 items scored from 0-3, with a higher score indicating more anxiety symptom
Brunnsviken Brief Quality of life scale | From enrollment to end of treament at 9 weeks. Follow-ups at 24 and 36 months after end of treatment.
  Measures quality of life. 12 items scored from 0-4. A higher score indicates higher quality of life

OTHER OUTCOMES:
Patient Health Questionnaire - 4 | From enrollment on a weekly basis through study completion 9 weeks later.
  Brief measurer of depressive and anxiety symptoms. Consists of 4 items, scored from 0-3. A higher score indicates more symptoms.
Client Satisfaction Questionnaire | At week 9 following enrollment.
  CSQ is used to assess client satisfaction with health and human services. Total scores range from. 8 to 32, with the higher number indicating greater satisfaction.
The Morisky Medication Adherence Scale | From enrollment to end of treament at 9 weeks.
  The Morisky Medication Adherence Scale (MMAS-8) is an 8-item structured, self-report measure that assesses medication adherence. Higher scores indicates higher adherence

CONTACTS AND LOCATIONS:
Locations (1):
- Linköping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared on request following initial publication of results.